CLINICAL TRIAL: NCT00452127
Title: An Open-Label, Multicenter, Phase I/II Trial of the Safety of Escalating Doses of PRO131921 in Patients With Relapsed or Refractory Indolent Non-Hodgkin's Lymphoma Who Have Been Treated With a Prior Rituximab-Containing Regimen
Brief Title: A Trial of the Safety of Escalating Doses of PRO131921 in Patients With Relapsed or Refractory Indolent Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACO3967g
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: NHL; Indolent; Follicular
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — PRO131921 monoclonal antibody

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PRO131921

INTERVENTIONS:
Drug: PRO131921 — Escalating doses by IV infusion

SUMMARY:
This is an open-label, multicenter, Phase I/II study of the safety of escalating doses of single-agent PRO131921 in patients with relapsed or refractory CD20-positive indolent NHL. The trial will enroll in two phases: a Phase I dose-escalation portion for patients with indolent NHL and a Phase II portion with enrollment of additional patients with follicular NHL into two expanded treatment cohorts in order to expand the safety database and collect preliminary anti-lymphoma activity data.

ELIGIBILITY:
* Signed informed consent
* Ability and willingness to comply with the requirements of the study protocol
* Age ≥ 18 years
* Documented history of histologically confirmed CD20-positive follicular NHL (Phases I and II); for Phase I, other CD20-positive indolent lymphomas (marginal zone lymphoma and small lymphocytic lymphoma) are also included. Patients with a history of a CD20-positive NHL of mixed (indolent/aggressive) histology may also be included in Phase I if the most recent relapse biopsy shows only indolent NHL
* Indolent lymphoma (Phase I) or follicular lymphoma (Phase II) that either has relapsed after a documented history of response (CR, CRu, or PR) of ≥6 months to a rituximab-containing regimen or was refractory to a previous rituximab-containing regimen
* Bi-dimensionally measurable disease, with at least one lesion >1.5 cm in its largest dimension
* Absolute B-cell count ≥LLN at screening (Phase I only)
* ECOG performance status of 0, 1, or 2
* For patients of reproductive potential (males and females), use of a reliable means of contraception during the study and for 1 year following the last dose of study treatment
* For females of childbearing potential, a negative serum pregnancy test within 14 days prior to enrollment

Exclusion Criteria:

* Prior use of anti-CD20 monoclonal antibody therapy (other than rituximab or radioimmunotherapy)
* Prior use of any non-CD20-targeted monoclonal antibody therapy within 6 months of enrollment
* Current or recent lymphoma treatment
* History of severe allergic or anaphylactic reactions to human, humanized, chimeric, or murine monoclonal antibodies
* Evidence of significant uncontrolled concomitant diseases, such as cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine, or gastrointestinal disorders
* Evidence of myelodysplasia or myelodysplastic changes on bone marrow examination
* Untreated or persistent/recurrent malignancy (other than lymphoma)
* Known active bacterial, viral, fungal, mycobacterial, or other infection
* A major episode of infection requiring hospitalization or treatment with IV antimicrobials within 4 weeks of screening or oral antimicrobials within 2 weeks of screening
* History of recurrent significant infection or bacterial infections
* Positive hepatitis B or C serology
* Positive human immunodeficiency virus (HIV) serology
* Pregnancy or lactation
* Central nervous system lymphoma
* Recent major surgery within 4 weeks of screening, other than diagnostic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-05; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities and adverse events | Length of study

SECONDARY OUTCOMES:
Pharmacokinetic parameters; CD19-positive B-cell counts | Length of study
Overall response; and progression-free survival (Ph. 2 only) | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Bill Ho, M.D., Study Director — Genentech, Inc.